CLINICAL TRIAL: NCT03586388
Title: Pilot Study on the Efficacy and Safety of an Oral Desensitization Protocol at the Onset of Food Allergy
Brief Title: Early Oral Immunotherapy in Infants With Cow's Milk Protein Allergy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC 18/12
Record Dates: First submitted 2018-07-02; First posted 2018-07-13 (Actual); Last update posted 2018-07-16 (Actual); Status verified 2018-07

CONDITIONS: Hypersensitivity, Milk
Keywords: Hypersensitivity, Milk; Cow's Milk; Immunotherapy; Infant
MeSH Terms: conditions — Milk Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oral immunotherapy protocol (Experimental): Eligible children receive the oral food challenge (OCD) protocol
  Interventions: Other: Oral immunotherapy protocol

INTERVENTIONS:
Other: Oral immunotherapy protocol — In hospital setting: three increasing doses every 30 minutes of 1ml, 5ml and 10ml of cow milk (CM). Oral food challenge (OFC) stopped at 10ml even if no clinical reactions occurred.
  At home: every child will take the dose tolerated in hospital, starting the day after the OFC, for 3-4 weeks.Once reached the dose of 40ml of CM without reactions for at least 2 weeks, families increment the dose of 5 ml every week, till the tolerance of 50 ml, then of 10 ml every week, till the tolerance of 100ml and then, of 10 ml every 3 days till the tolerance of 150 ml of milk.
  Other Names: Oral food challenge (OCD)

SUMMARY:
Cow's milk (CM) allergy is the most frequent food allergy in the first years of life, with prevalence rates estimated in the range of 2-3%.

The elimination of CM is the mainstay of treatment, but accidental exposure to CM proteins is not uncommon, with a considerable risk of severe allergic reactions.

Recent evidence suggests that early oral exposure in young children may protect to the development of allergy. On the same way, strategies have been developed for the use of oral exposure as immunotherapy for the treatment of children with established food allergy even if available data on the use of oral immunotherapy in infants with food allergy are very limited.

The aim of this study is to evaluate the feasibility of an oral immunotherapy protocol, started in the first year of life, in children with CM allergy.

ELIGIBILITY:
Inclusion Criteria:

• children between 3-12 months with CM allergy (defined as the association of typical clinical manifestations in the first hour after CM ingestion and evidence of sensitization of CM proteins on both skin prick test and specific serum IgE levels)

Exclusion Criteria:

* children with not IgE-mediated clinical manifestations
* children with a known immunodeficiency

Ages: 3 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 73 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
number of children that completed the home oral immunotherapy protocol, reaching clinical tolerance | 6 months
  Clinical tolerance defined as the achievement of a dose of 150 ml of CM or a corresponding dose of dairy products

SECONDARY OUTCOMES:
Clinical reactions experienced by children at home | 6 months
  Number and types, communicated by parents at a dedicated telephone number.
Serum levels of specific IgE | 6 months
  Comparison in serum levels of specific IgE between baseline and the end of the protocol, hypothesizing a decrease of IgE levels after OFC
Serum levels of specific IgG4 | 6 months
  Comparison in serum levels of specific IgG4 between baseline and the end of the protocol, hypothesizing an increase of IgG4 levels after OFC

CONTACTS AND LOCATIONS:
Overall Officials: Laura Badina, Md, Principal Investigator — IRCCS Burlo Garofolo; Giorgio Longo, MD, Study Chair — IRCCS Burlo Garofolo; Egidio Barbi, MD, Study Director — IRCCS Burlo Garofolo
Locations (1):
- Institute for Maternal and Child Health - IRCCS Burlo Garofolo-, Trieste, Italy